CLINICAL TRIAL: NCT05105854
Title: Hand Osteoarthritis: Investigating Pain Trajectories and Association With Biomarkers Including Estrogen Cohort
Acronym: HOPE-c
Status: Active, not recruiting | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: Versus Arthritis (Other)
Responsible Party: Sponsor
Other Study IDs: 14602
Record Dates: First submitted 2021-10-22; First posted 2021-11-03 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-10

CONDITIONS: Hand Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Adults with painful hand osteoarthritis are invited to take part in this observational cohort study. The course of hand pain can vary and is not well understood - some people seem to have short episodes of worsening pain ('flares') and the trend (or 'trajectory') over a longer period of time may be of improvement, staying stable or worsening. The study aims to identify and define different pain trajectories in hand OA, including factors which may predict the future course of pain in the condition.

Due to the Covid-19 pandemic, currently all study related activities are being carried out remotely (online, by post, by phone).

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent to participate in the study.
* Aged 18 years or above
* The participant reports a diagnosis of hand osteoarthritis made by a health care professional OR (Optional inclusion, for review after 3 months*) The participant reports a diagnosis of hand osteoarthritis

  * Given the Covid-19 pandemic, it is not clear if requiring a health care professional diagnosis will limit participation in the study. If, after 3 months of recruitment, fewer than 24 participants have been recruited, self-reported diagnosis, supported by additional materials available on the study website or by discussion with a study team member by phone will be acceptable. Numbers in each of these two categories will be recorded.
* Two or more painful hand joints: interphalangeal and/or base of thumb
* Hand pain on most days of the last month i.e. ≥15 days in the last month
* Competency of English language that permits written informed consent and independent completion of questionnaires

Exclusion Criteria:

The participant may not enter the study if any of the following apply:

* Other cause for hand pain including rheumatoid arthritis, psoriatic arthritis, gout, haemochromatosis or connective tissue disease.
* Current or previous diagnosis of psoriasis
* Any additional condition which is substantially contributing to hand pain or would confound the measurement of hand pain, including but not limited to: chronic widespread pain, active tenosynovitis causing hand pain, active carpal tunnel syndrome, active cervical radiculopathy
* Recent change in treatments

  * Within the last four weeks:

Initiation of new analgesic or change in usual dose or route; Use of oral steroids or intraarticular steroid to sites other than the hand

* Within the last three months:

Use of intraarticular steroid to the hand; Initiation of glucosamine, chondroitin, hand exercises or other relevant non- pharmacological therapy for hand pain; Initiation or change in dose, route or formulation of hormonal therapy (such as hormone replacement or contraceptive); Use of intramuscular steroid

* Within the last six months:

Use of immunosuppressive treatment; Hand surgery within the last six months, or planned within the next six months; Use of intra-articular hyaluronan to the hand in the last six months

* Current participant in an interventional research trial that involves blinding of treatment allocation
* Any other significant or uncontrolled disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with painful hand osteoarthritis
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-07-07 (Actual); Primary Completion 2029-02-07 (Estimated); Study Completion 2029-02-07 (Estimated)

PRIMARY OUTCOMES:
To identify and define different pain trajectories in hand OA. | 6 months
  Average hand pain (daily rating)

SECONDARY OUTCOMES:
To identify predictors of pain trajectories in hand OA. | 6 months
  Trajectory Category (as determined by the primary objective), which may include persistent stable, persistent worsening, resolving, fluctuating, presence of flares
To test whether there is an association between changes in sex hormone levels and hand pain severity over time within an individual | The previous 7 days and for 7 days after the study visit, up to 6 months
  Hand pain (0 to 10 on a numerical rating scale)
To identify whether pre-defined variables are: a) Baseline predictors of flare/change during the study b) Associated with the presence of flare/change in hand symptoms | 6 months, 2 years 5 years
  Presence of flare/change in hand pain (yes/no) as self-reported by the participant
To characterise features of a flare in hand OA | At time of self reported flare (the previous 7 days and for 7 days after the study visit)
  Clinical history (antecedent events, sleep quality and disturbance, analgesic use); Pain measures: to identify a numerical definition (0-10 on NRS) of pain flare in hand OA; Duration of a flare; Morning stiffness (minutes); Clinical examination including Grip Strength; Hand Function (Functional Index for Hand Osteoarthritis (FIHOA) Questionnaire); Brief Pain Inventory Short Form; Global Well-being Visual Analogue Scale (0-100); Hospital Anxiety and Depression Scale (HADS); Anger/Frustration Short Form questionnaire (PROMIS); Features on hand photograph; Acoustic emission from hand movements
To assess the following optional features: a) Use of local daily weather recordings and study its association with daily hand pain rating b) Identification of any acoustic emissions that are associated with features of hand OA | 6 months
  Daily weather recording, derived from a Meteorological Service website (including temperature, pressure, humidity, precipitation, wind speed)
  Acoustic emissions from hand movements

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Charing Cross Hospital, Imperial College Healthcare NHS Trust, London
  - Nuffield Orthopaedic Centre, Oxford University Hospitals NHS Foundation Trust, Oxford

IPD SHARING:
Plan to Share IPD: Undecided
No data sharing policy established as yet. Potential collaborators may contact the Chief Investigator relating to bone fide research proposals.

REFERENCES:
- See also: This link will take you to the study website which contains more information about the study as well as information about how to take part. — http://www.hopecohort.org.uk